CLINICAL TRIAL: NCT04180072
Title: Atezolizumab Plus Bevacizumab for Patients With Advanced Hepatocellular Carcinoma (HCC) and Chronic Hepatitis B Virus (HBV) Infection
Brief Title: Atezolizumab Plus Bevacizumab With HCC and HBV Infection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Changhua Christian Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2219
Record Dates: First submitted 2019-11-24; First posted 2019-11-27 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab plus bevacizumab (Experimental): Atezolizumab 1200 mg IV plus bevacizumab 15 mg/kg IV on day 1 every 3 weeks. Study treatment will continue until documented tumor progression or occurrence of unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg IV on day 1 every 3 weeks
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab 15 mg/kg IV on day 1 every 3 weeks
  Other Names: Avastin

SUMMARY:
This is a single-arm clinical trial. The main objective is to determine the efficacy of atezolizumab+bevacizumab therapy in patients with advanced hepatocellular carcinoma and with chronic hepatitis B virus infection. All eligible patients will receive atezolizumab + bevacizumab therapy.

DETAILED DESCRIPTION:
Combination of atezolizumab, an immune checkpoint inhibitors (ICI), and bevacizumab, an anti-angiogenic antibody, has shown promising anti-tumor activity and good safety profile in patients with advanced hepatocellular carcinoma (HCC) and good liver function reserves (Child-Pugh class A). Currently all trials of ICI-based therapy for HCC enrolled only patients with very low HBV viral loads if they had chronic HBV infection because of the concern of the risk of HBV reactivation on the severity and management of liver-related adverse events, particularly immune-related hepatitis.

The investigators hypothesize that in patients with advanced HCC, chronic HBV infection, and adequate liver function reserves, the safety profile of ICI-based therapy should be similar to those in other patient populations as long as prophylactic anti-HBV treatment is given, regardless the baseline HBV viral load. This is because in patients with patients with lymphoma and chronic HBV infection, who have the highest risk of HBV reactivation after cytotoxic or immunosuppressive therapy, no HBV-related complications of clinical significance were noted as long as prophylactic anti-HBV treatment started before the administration of cytotoxic or immunosuppressive therapy.

This is a single-arm clinical trial. Key eligibility criteria will include the following: histologically proven, locally advanced or metastatic and/or unresectable HCC that is not amenable to curative surgical and/or locoregional therapies; no prior systemic therapy for HCC; documented chronic HBV infection with HBV DNA > 2000 IU/mL obtained within 28 days prior to initiation of study treatment; at least one measurable (per RECIST 1.1) lesion; ECOG Performance Status of 0 or 1; and Child-Pugh class A.

All eligible patients will receive atezolizumab 1200 mg IV plus bevacizumab 15 mg/kg IV on day 1 every 3 weeks. Study treatment will continue until documented tumor progression or occurrence of unacceptable toxicity. All eligible subjects will receive anti-HBV treatment (per local standard of care; e.g., entecavir) prior to start of study treatment and continue anti-HBV treatment for the length of the study. The primary endpoint is overall response rate defined as a complete or partial response, as determined by the investigator according to RECIST v1.1. The secondary endpoints will include safety measures (e.g., the proportion of subjects with ≥ grade 3 liver-related adverse events (AE) (according to NCI CTCAE v5.0), incidence and severity of all adverse events/ immune-related adverse events, incidence of HBV reactivation/ HBV-related hepatitis flare) and efficacy measures (e.g., objective response rate, progression-free survival, duration of response, and overall survival). This study plan to enroll 48 evaluable subjects, defined as subjects who receive 3 cycles of study treatment and the first image evaluation for tumor response. The estimated time of enrollment will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years, according to local regulation in Taiwan, at time of signing Informed Consent Form.
* Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology.
* Agreement to receive a mandatory tumor biopsy for enrollment into this study.
* Disease that is not amenable to curative surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies.
* No prior systemic therapy (including systemic investigational agents) for HCC.
* Documented chronic HBV infection, defined by positive serum surface antigen (HBsAg), and HBV DNA > 2000 IU/mL obtained within 28 days prior to initiation of study treatment.
* Agreement to receive anti-HBV treatment (per local standard of care; e.g., entecavir)

  1 to 2 weeks prior to study entry and willingness to continue treatment for the length of the study.
* At least one measurable (per RECIST 1.1) lesion. Patients who received prior local therapy (e.g., radiofrequency ablation or transarterial chemoembolization, etc.) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST version 1.1.
* ECOG Performance Status of 0 or 1 within 7 days prior to registration.
* Child-Pugh class A (see Appendix) within 14 days prior to registration
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 7 days prior to registration, unless otherwise specified:

  * ANC ≥ 1.5 x 109/L (1500/μL) without granulocyte colony-stimulating factor support; platelet count ≥ 75 x 109/L (75,000/μL) without transfusion; and hemoglobin ≥ 90 g/L (9 g/dL)(patients may be transfused to meet this criterion).
  * Liver transaminases (AST and ALT) ≤ 5 x upper limit of normal (ULN)
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
  * Urine dipstick for proteinuria < 2+ (within 7 days prior to initiation of study treatment).

Patients who have ≥ 2+ proteinuria on dipstick urinalysis at baseline will be eligible if he/she have daily protein excretion of < 1 g documented by a 24-hour urine collection.

* Women of childbearing potential must agree to use contraceptive methods with a failure rate of < 1% per year (e.g., hormonal contraceptives that inhibit ovulation, copper intrauterine devices) during the treatment period and for at least 5 months after the last dose of atezolizumab, and 6 months after the last dose of bevacizumab.
* Men must agree to use contraceptive measures (condom plus an additional contraceptive method that together result in a failure rate of < 1% per year) during the treatment period and for 6 months after the last dose of bevacizumab.

Exclusion Criteria:

* Histological diagnosis of fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Imaging finding for HCC corresponding to any of the following:

  o Clear invasion into the bile duct
* Co-infection of HBV and HCV. Patients with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV.
* Known human immunodeficiency virus (HIV) infection.
* History of esophageal/gastric varices or active peptic ulcers that are considered to have high risk of bleeding.
* History of upper gastrointestinal bleeding within 1 year.
* Major systemic diseases that the investigator considers inappropriate for participation.
* History of severe allergic anaphylactic reactions to antibodies or fusion proteins
* Prior allogeneic stem cell or solid organ transplantation.
* Treatment with investigational therapy within 28 days prior to initiation of study treatment.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* Local therapy to liver (e.g., radiofrequency ablation, transarterial chemoembolization, etc.) within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure.
* Radiotherapy within 28 days and abdominal/ pelvic radiotherapy within 60 days prior to initiation of study treatment, except for palliative radiotherapy to bone lesions.

Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.

* Presence of central nervous system (CNS) or leptomeningeal metastases. Patients with a history of CNS metastases are eligible for the study if he/she have received radiotherapy or surgery for the CNS metastases, and complete response (no evidence of residual CNS metastases) must be documented by brain CT scan at screening.
* Any active autoimmune disease or history of known autoimmune disease except for vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* History of drug-induced pneumonitis or idiopathic pneumonitis, or Evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Known active tuberculosis or other active infection.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment. Core biopsy or other minor surgical procedure within 3 days prior to the first dose of bevacizumab
* History of malignancy other than HCC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer.
* Requirement of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) ≥150 mmHg and/or diastolic blood pressure > 100 mmHg), based on an average of ≥ 3 BP readings on ≥ 2 sessions, despite optimal antihypertensive therapy..
* Current or recent (within 10 days of first dose of study treatment) use of aspirin (> 325 mg/day), other anti-platelet therapy (e.g., dipyramidole, ticlopidine, clopidogrel, and cilostazol), or full dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa) and rivaroxaban (Xarelto) is not recommended due to bleeding risk.
* History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment), unstable arrhythmia, or unstable angina
* History of uncorrectable electrolyte disorder affecting serum levels of potassium, calcium, or magnesium
* Treatment of active infection with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the last dose of atezolizumab
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulation
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding .Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of study treatment do not need to repeat the procedure.
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
* Moderate or severe ascites
* History of hepatic encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of hemoptysis (≥2.5 mL of bright red blood per episode) within 1 month prior to initiation of study treatment
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fractureMetastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses (<30 mm from the carina) of large volume Patients with vascular invasion of the portal or hepatic veins may be enrolled.
* History of intra-abdominal inflammatory process within 6 months prior to initiation of study treatment, including but not limited to active peptic ulcer disease, diverticulitis, or colitis
* Uncontrolled tumor-related pain Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurX) are allowed.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor approval has been obtained. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Best overall response rate | The last patient in has been treated for 6 months. All patients who have a PR or CR before that are responders
  Complete or partial response, as determined by the investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Proportion of subjects with ≥ grade 3 liver-related adverse events (AE) | 12 weeks after the first drug administration.
  Proportion of subjects with ≥ grade 3 liver-related adverse events (AE) according to NCI CTCAE v5.0
Incidence and severity of total AE, liver related AE, and liver immune-related AE | 30 days after the last dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurs first
  Any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment
HBV reactivation | Baseline up to approximately 2.5years.
  (1) HBV DNA increase of ≧ 100 folds than baseline level, regardless of alanine aminotransferase (ALT) changes; (2) HBV DNA increase of ≧ 10 folds than baseline level, associated with significant ALT changes (defined as ≧ 3-fold increase in ALT, compared with baseline levels, and increase in ≧ 1 grade defined by CTCAE5.0); and (3) 2 consecutive increase in HBV DNA of ≧ 100 folds than previous nadir level, regardless of ALT changes.
HBV-related hepatitis flare | Every 4 weeks for 6 months in permanent discontinuation of study drug treatment
  HBV reactivation plus ≧ 3-fold increase in alanine aminotransferase (ALT), compared with baseline levels, and increase in ≧ 1 grade defined by CTCAE v 5.0
Progression-free survival | The time from registration to the first occurrence of disease progression or death from any cause (whichever occurs first assessed up to 100 months)
  The time from registration to the first occurrence of disease progression or death from any cause (whichever occurs first)
Time to tumor progression | The time from registration to the first occurrence of disease progression assessed up to 100 months
  The time from registration to the first occurrence of disease progression
Duration of response | The time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first assessed up to 100 months)
  The time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first)
Disease stabilization rate | Complete response + partial response + stable disease lasting for ≧16 weeks approximately1years.
  Complete response + partial response + stable disease lasting for ≧16 weeks
AFP response | 9 weeks ± 1 week after the first drug administration
  ≥ 20% decrease from baseline at the first response assessment
Overall survival | The time from registration to death from any cause assessed up to 100 months
  The time from registration to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Chiun Hsu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (7):
- Taiwan (7):
  - Chang Gung Memorial Hospital, Linkou District
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No